CLINICAL TRIAL: NCT01135420
Title: Dual Diagnosis Inpatients: Telephone Monitoring RCT to Improve Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IAC 09-055
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Diagnosis, Dual (Psychiatry)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Psychiatry inpatient usual care
  Interventions: Other: Usual care
- Telephone Monitoring (Experimental): Patients in the TM condition will receive an in-person session while in treatment, followed by monitoring over the telephone for three months after discharge. The intervention will incorporate motivational interviewing to monitor patients' substance use, facilitate entry into outpatient treatment, and encourage 12-step self-help group participation.
  Interventions: Behavioral: Telephone Monitoring (TM) with Motivational Interviewing

INTERVENTIONS:
Behavioral: Telephone Monitoring (TM) with Motivational Interviewing — Patients in the TM condition will receive an in-person session while in the inpatient psychiatry program, followed by monitoring delivered over the telephone for three months after discharge. The TM intervention will have a motivational interviewing component to address patients' motivation to obtain help for and reduce their substance abuse. The purpose of the intervention condition is to monitor patients' substance use, facilitate patients' entry into outpatient substance use disorder (SUD) treatment, and encourage ongoing 12-step selfhelp group participation to support sobriety.
  Arms: Telephone Monitoring
Other: Usual care — All patients in the trial will receive usual care (i.e., the care they would have received in the absence of a study).
  Arms: Usual Care

SUMMARY:
This research program will improve the care and treatment outcomes of dually diagnosed veterans who receive inpatient psychiatry care, and decrease their use of VA inpatient mental health services. It will increase the use of substance abuse outpatient care and 12-step groups to benefit recovery, reduce rehospitalizations, and reduce costs for VA.

DETAILED DESCRIPTION:
Background:

Substance use disorders (SUDs) are highly prevalent among veteran psychiatry inpatients. Dual substance use and psychiatric disorders are related to poor outcomes and rehospitalizations, which are quite costly. However, relatively little is known about how to effectively help dually diagnosed psychiatry inpatients. Telephone Monitoring (TM) is effective among SUD patients at increasing SUD continuing care and self-help utilization and improving SUD outcomes. This study will build on these findings and contribute important new clinical knowledge by determining whether TM is similarly effective when adapted for dually diagnosed veteran psychiatry inpatients. It will evaluate the effectiveness of a manual-guided TM intervention.

Objectives:

Primary hypotheses are that patients in the TM condition, compared to patients in usual care (UC), will attend more SUD continuing care sessions and 12-step group meetings, and have better SUD and psychiatric outcomes. Secondary hypotheses are that TM patients will have fewer and delayed rehospitalizations, and their better outcomes will be mediated by SUD outpatient treatment and 12-step group participation.

Methods:

This study will take place at two VAs: Palo Alto (VISN 21) and Ann Arbor (VISN 11). Dually diagnosed patients in psychiatry inpatient treatment will be randomly assigned to UC or TM. Patients in the TM condition will receive an in-person session while in treatment, followed by monitoring over the telephone for three months after discharge. The intervention will incorporate motivational interviewing to monitor patients' substance use, facilitate entry into outpatient treatment if a relapse occurs, and encourage 12-step self-help group participation. Patients will be assessed at baseline, end-of-intervention, and six months and one-year post-intervention for primary and secondary outcomes and non-VA health care; VA health care will be assessed with VA databases. GLMM analyses will be conducted to compare the UC and TM groups on course of primary and secondary outcomes over time; Cox regression models will compare groups on time to rehospitalization; and sequential regression analyses will examine whether outcomes associated with TM are mediated by more SUD continuing care and 12-step group participation.

Status:

As of this time, this project is in the follow-up data collection phase.

ELIGIBILITY:
Inclusion Criteria:

* Dually diagnosed veteran in VA inpatient psychiatry treatment

Exclusion Criteria:

* Current diagnosis of schizophrenia or schizoaffective disorder
* too psychiatrically unstable or cognitively impaired to understand informed consent and other study procedures
* does not have ongoing telephone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

REFERENCES:
- [Result] Timko C, Cronkite RC, McKellar J, Zemore S, Moos RH. Dually diagnosed patients' benefits of mutual-help groups and the role of social anxiety. J Subst Abuse Treat. 2013 Feb;44(2):216-23. doi: 10.1016/j.jsat.2012.05.007. Epub 2012 Jul 3. PMID 22763197
- [Result] Timko C, Bonn-Miller MO, McKellar JD, Ilgen MA. Detoxification history and two-year outcomes of substance use disorder treatment and mutual-help group participation. Journal of drug issues. 2014 Jan 1; 44(1):4-21.
- [Result] Woodhead E, Cowden Hindash A, Timko C. Dual Diagnosis, Mutual-Help Use, and Outcomes: A Naturalistic Follow-Up. Journal of Dual Diagnosis. 2013 May 3; 9(2):158-164.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from inpatient psychiatry settings.
Groups:
- Usual Care: Psychiatry inpatient usual care
  Usual care: All patients in the trial received usual care (i.e., the care they would have received in the absence of a study).
- Telephone Monitoring: Patients in the TM condition received an in-person session while in treatment, followed by monitoring over the telephone for three months after discharge. The intervention incorporated motivational interviewing to monitor patients' substance use, facilitate entry into outpatient treatment, and encourage 12-step self-help group participation.
  Telephone Monitoring (TM) with Motivational Interviewing: Patients in the TM condition received an in-person session while in the inpatient psychiatry program, followed by monitoring delivered over the telephone for three months after discharge. The TM intervention had a motivational interviewing component to address patients' motivation to obtain help for and reduce their substance abuse. The purpose of the intervention condition was to monitor patients' substance use, facilitate patients' entry into outpatient substance use disorder (SUD) treatment, and encourage ongoing 12-step selfhelp group participation to support sobriety.
Period: Overall Study
Arm/Group | Usual Care | Telephone Monitoring
Started | 199 | 207
Completed | 155 | 175
Not Completed | 44 | 32

BASELINE CHARACTERISTICS:
Groups:
- Telephone Monitoring: Patients in the TM condition received an in-person session while in treatment, followed by monitoring over the telephone for three months after discharge. The intervention will incorporate motivational interviewing to monitor patients' substance use, facilitate entry into outpatient treatment, and encourage 12-step self-help group participation.
  Telephone Monitoring (TM) with Motivational Interviewing: Patients in the TM condition will receive an in-person session while in the inpatient psychiatry program, followed by monitoring delivered over the telephone for three months after discharge. The TM intervention will have a motivational interviewing component to address patients' motivation to obtain help for and reduce their substance abuse. The purpose of the intervention condition is to monitor patients' substance use, facilitate patients' entry into outpatient substance use disorder (SUD) treatment, and encourage ongoing 12-step selfhelp group participation to support sobriety
- Total: Total of all reporting groups
Arm/Group | Usual Care | Telephone Monitoring | Total
Number analyzed (Participants) | 199 | 207 | 406
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (13) | 45 (13) | 45 (13)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 183 | 189 | 372
Region of Enrollment [Number; unit: participants]
  United States | 199 | 207 | 406

OUTCOME MEASURES:

1. Primary Outcome: Readiness to Attend Substance Use Disorder Continuing Care
Description: Readiness to attend substance use disorder continuing care; scale range=0-4, with 0=not ready to do; 4=already doing; higher scores indicate a better outcome.
Time Frame: 3 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Telephone Monitoring
Number analyzed (Participants) | 155 | 175
units on a scale | 1.8 (1.1) | 2.2 (1.3)
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority or Other; p < .05, ANCOVA; Mean Difference (Final Values) = 0.4

ADVERSE EVENTS:
Arm/Group | Usual Care | Telephone Monitoring
Serious Adverse Events (participants affected / at risk) | 3/199 | 4/207
Other Adverse Events (participants affected / at risk) | 3/199 | 4/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=199) | Telephone Monitoring (N=207)
death (Cardiac disorders) | 3 | 4 — This is death from cardiac-related causes.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=199) | Telephone Monitoring (N=207)
hospitalization (Psychiatric disorders) | 3 (3) | 4 (4) — No additional description

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes